CLINICAL TRIAL: NCT04647812
Title: Technology-assisted Rehabilitation After Acute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vetrea Terveys Oy (Other)
Collaborators: Kuopio University Hospital (Other); City of Kuopio (Other Government)
Responsible Party: Principal Investigator, Kauko Pitkänen, Chief physician, Vetrea Terveys Oy
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Taku2020
Record Dates: First submitted 2020-11-30; First posted 2020-12-01 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Consecutive cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Technology-assisted rehabilitation (Experimental): Augmented exercise therapy with novel technology
  Interventions: Behavioral: Technology-assisted rehabilitation
- Conventional rehabilitation (Experimental): Traditional multidisciplinary rehabilitation
  Interventions: Behavioral: Conventional rehabilitation

INTERVENTIONS:
Behavioral: Technology-assisted rehabilitation — Augmented exercise therapy with novel technology and home-based telerehabilitation
  Arms: Technology-assisted rehabilitation
Behavioral: Conventional rehabilitation — Traditional multidisciplinary in-patient rehabilitation
  Arms: Conventional rehabilitation

SUMMARY:
The aim of the study is to evaluate the effects and costs of an intensified rehabilitation for stroke patients. Using novel technologies the patients will receive an augmented exercise therapy during the first weeks after stroke. The effects on restoration of functions as well as on the costs incurred from social and health care services will be assessed and compared to the conventional rehabilitation over 6 month follow-up.

DETAILED DESCRIPTION:
The intervention consists of technology-assisted multidisciplinary rehabilitation for 3 weeks followed by an 8-week period of supervised home-based telerehabilitation and a weekly group exercise in an outpatient clinic. The effects on mobility, upper extremity motor functions and activities of daily living will be assessed using FAC, hand grip force, shoulder elevation test, WHODAS 2.0 and PROMIS scales. The costs incurred from social and health care services over 6 months will be compared to the control group receiving conventional rehabilitation. Patients aged 18 or more with their first stroke and stable cardiopulmonary condition will be consecutively recruited first into the control group (n=20) and thereafter into the experimental group (n=20). Patients with a severe cognitive deficit or aphasia will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or more
* first stroke

Exclusion Criteria:

* unstable cardiopulmonary condition
* severe cognitive disorder
* aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
WHODAS 2.0 | 6 months
  World Health Organization Disability Assessment Schedule - 12 questions scoring 1 to 5 yielding a total score from 12 to 60. A higher score means an increasing disability.
service use and costs | 6 months
  amount and costs of social and health care services used

SECONDARY OUTCOMES:
PROMIS Global 10 | 6 months
  Patient Reported Outcome Measurement Information System - a generic global health scale v1.2 consists of 10 questions across 6 health items. Two of the items (Physical and Mental) can be converted to T-scores allowing comparisons to a general population.
FAC | 6 months
  Functional Ambulation Categories - categorical scale ranging from 0 (unable to walk) to 5 (independent walking without assistive devices on any surfaces).
Hand grip force | 6 months
  hand grip
Shoulder elevation test | 6 months
  shoulder range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Kauko Pitkänen, MD, PhD, Study Director — Vetrea Terveys Oy
Locations (1):
- Vetrea, Kuopio, Northern Savonia, Finland